CLINICAL TRIAL: NCT01279265
Title: Effect of Lactobacillus Rhamnosus GG (LGG) on Infant Crying, Intestinal Microbiota, and Intestinal Inflammation in Infants With Colic
Brief Title: Effect of Lactobacillus Rhamnosus GG (LGG) on Infant Colic
Acronym: LGG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Mead Johnson Nutrition (Industry)
Responsible Party: Principal Investigator, J. Marc Rhoads, Professor - Pediatrics, Gastroenterology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HSC-MS-10-0048
Record Dates: First submitted 2011-01-12; First posted 2011-01-19 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Colic; Inflammation
Keywords: Lactobacillus; Probiotic; Crying time; Fecal microbiota; Calprotectin; Colic; Infant Crying; Barr Diary; Breath Hydrogen; Clinical Design
MeSH Terms: conditions — Colic; Inflammation | interventions — pregestimil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutramigen Lipil with Enflora (Active Comparator): Formula with probiotics (Lactobaccillus Rhamnosus GG)
  Interventions: Dietary Supplement: Nutramigen with Enflora
- Nutramigen A+ (Placebo Comparator): Hypoallergenic formula without probiotics (Lactobaccillus Rhamnosus GG)
  Interventions: Dietary Supplement: Nutramigen A+

INTERVENTIONS:
Dietary Supplement: Nutramigen with Enflora — Hypoallergenic formula with probiotic - Lactobacillus GG
  Arms: Nutramigen Lipil with Enflora
Dietary Supplement: Nutramigen A+ — Hypoallergenic formula without lactobacillus
  Other Names: (Nutramigen Lipil)
  Arms: Nutramigen A+

SUMMARY:
This study will compare 2 currently marketed formulas in healthy full term babies: Nutramigen A+ (a hypoallergenic formula) and Nutramigen-Enflora (hypoallergenic formula with Lactobacillus GG (LGG)) during 3 months of formula feeding. The investigators' aims are to compare 3 outcomes in these babies: (1) normal baby crying time; (2) the composition of intestinal microbiota (bacteria in the stool); and (3) a lab test which measures the number of white blood cells in the large intestine (fecal calprotectin). The investigators predict that LGG supplementation (Nutramigen-Enflora) will facilitate its establishment as an important component of the neonatal intestinal microbial community and reduce fecal calprotectin.

ELIGIBILITY:
Inclusion Criteria:

* Sixty healthy full-term colicky infants (gestational age 32 wks to 41 wks)

Exclusion Criteria:

* chronic lung disease,
* diarrhea (stools that take the shape of a container > 5x daily)
* fever

Ages: 3 Weeks to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. M Rhoads, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Background] Rhoads JM, Fatheree NY, Norori J, Liu Y, Lucke JF, Tyson JE, Ferris MJ. Altered fecal microflora and increased fecal calprotectin in infants with colic. J Pediatr. 2009 Dec;155(6):823-828.e1. doi: 10.1016/j.jpeds.2009.05.012. Epub 2009 Jul 22. PMID 19628216
- [Derived] Rhoads JM, Collins J, Fatheree NY, Hashmi SS, Taylor CM, Luo M, Hoang TK, Gleason WA, Van Arsdall MR, Navarro F, Liu Y. Infant Colic Represents Gut Inflammation and Dysbiosis. J Pediatr. 2018 Dec;203:55-61.e3. doi: 10.1016/j.jpeds.2018.07.042. Epub 2018 Aug 31. PMID 30177353

RESULTS

PARTICIPANT FLOW:
Groups:
- Nutramigen A+: Hypoallergenic formula without lactobacilli
  Nutramigen A+: Hypoallergenic formula without lactobacillus
Period: Overall Study
Arm/Group | Nutramigen Lipil With Enflora | Nutramigen A+
Started | 13 | 17
Completed | 9 | 11
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nutramigen Lipil With Enflora | Nutramigen A+ | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 11 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Daily Average Crying and Fussing Duration According to Barr Diary Records
Description: The parent or guardian will complete a Barr diary to measure crying and fussing times of colicky infants . It is a daily timeline that records the number of minutes in five minute increments with fussiness and crying. The average colicky infant cries and fusses is more than 3 hours daily. If infants surpasses the 3 hours for more than three days (not consecutive) and are less than 3 months of age, they are considered to have colic.
Time Frame: 90 days
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Nutramigen Lipil With Enflora | Nutramigen A+
Number analyzed (Participants) | 9 | 11
minutes | 111 [65 to 157] | 133 [60 to 205]

2. Secondary Outcome: Fecal Microbiota
Description: Analyze and identify bacteria in the stool of the subjects. We will use pyrosequencing to characterize the bacteria colonizing the stool. We will measure diversity by Shannon's diversity index in the two groups.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Shannon's diversity index value
Arm/Group | Nutramigen Lipil With Enflora | Nutramigen A+
Number analyzed (Participants) | 9 | 11
Shannon's diversity index value
  Visit 1 - Baseline | .946 (.927) | .991 (.415)
  Visit 2- Day 14 | 1.314 (.789) | .537 (.289)
  Visit 3 - Day 42 | 1.047 (.350) | 1.161 (.612)
  Visit 4 - Day 90 | .676 (.444) | .737 (.409)

3. Secondary Outcome: Fecal Calprotectin
Description: Test intestinal inflammation in the infants. Calprotectin is made by white blood cells called neutrophils. The number of neutrophils in the intestine is reflected by the fecal calprotectin level.
Time Frame: 90 days
Measure: Mean (95% Confidence Interval); unit: µg/g (feces)
Arm/Group | Nutramigen Lipil With Enflora | Nutramigen A+
Number analyzed (Participants) | 9 | 11
µg/g (feces)
  Visit 1- Baseline | 285 [199 to 371] | 294 [184 to 404]
  Visit 2 - Day 14 | 226 [182 to 270] | 305 [186 to 423]
  Visit 3 - Day 42 | 229 [113 to 345] | 250 [154 to 347]
  Visit 4 - Day 90 | 211 [80 to 342] | 332 [225 to 440]

ADVERSE EVENTS:
Time Frame: 90 days (3 months)
Arm/Group | Nutramigen Lipil With Enflora | Nutramigen A+
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

LIMITATIONS AND CAVEATS:
75% of eligible babies either declined to enter the study or dropped out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No